CLINICAL TRIAL: NCT04744129
Title: NN414's Effect in Cerebral Hemodynamics and Headache Induction in Migraine Patients
Brief Title: Headache Inducing Effect of NN414 in Migraine Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Lili Kokoti, MD, PhD student, Principal investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: H-20009266
Record Dates: First submitted 2020-07-21; First posted 2021-02-08 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Headache, Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NN414 (Active Comparator): To investigate the role of NN414 compared with placebo in migraine patients.
  Interventions: Drug: NN414
- Saline (Placebo Comparator): To investigate the role of NN414 compared with placebo in migraine patients.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: NN414 — To investigate the role of NN414 on cerebral hemodynamic in migraine patients
  Other Names: 6-Chloro-3-[[1-methylcyclopropyl]amino]-4H-thieno[3,2-e]-1,2,4-thiadiazine 1,1-dioxide
  Arms: NN414
Drug: Saline — To investigate the role of NN414 compared with saline cerebral hemodynamic in migraine patients.
  Arms: Saline

SUMMARY:
To investigate the role of KATP channels on the cerebral hemodynamic in migraine patients.

ELIGIBILITY:
Criteria

Inclusion Criteria:

* Migraine patients of both sexes.
* 18-60 years.
* 50-100 kg.
* Women of childbearing potential must use adequate contraception.

Exclusion Criteria:

* Headache less than 48 hours before the tests start
* Daily consumption of drugs of any kind other than oral contraceptives
* Pregnant or nursing women.
* Cardiovascular disease of any kind, including cerebrovascular diseases.
* Diabetes mellitus and other endocrinologic disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Occurrence and change of migraine attack | Before (-10 min) and after infusion (+2 hours) of NN414 compared with before and after infusion of saline
  Occurrence of migraine according to international criteria

SECONDARY OUTCOMES:
Change in cerebral hemodynamic | Before (-10 min) and after infusion (+2 hours) of NN414 compared with before and after infusion of saline
  Change on velocity of media cerebri artery.
Occurrence and change of headache | Before (-10 min) and after infusion (+2 hours) of NN414 compared with before and after infusion of saline
  Occurrence of headache measured by numerical rating scale (NRS)
Change of diameter of the artery | Before (-10 min) and after infusion (+2 hours) of NN414 compared with before and after infusion of saline
  Change of diameter of superficial temporal artery and radial artery. The diameter will be measured by millimeter (mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Copenhagen, Capital Region, Denmark

REFERENCES:
- [Derived] Kokoti L, Al-Karagholi MA, Zhuang ZA, Amirguliyev S, Amin FM, Ashina M. Non-vascular ATP-sensitive potassium channel activation does not trigger migraine attacks: A randomized clinical trial. Cephalalgia. 2024 May;44(5):3331024241248211. doi: 10.1177/03331024241248211. PMID 38729773